CLINICAL TRIAL: NCT02139566
Title: Improving Consent and Survey Procedures for Young MSM in Web-based HIV Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Patrick S Sullivan, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IRB00065333; 1R21HD074502-01A1 (NIH)
Record Dates: First submitted 2014-05-11; First posted 2014-05-15 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Hi-tech video consent (Experimental): This group will be shown a professionally animated video that presents the major components of the informed consent document. Intervention is Video Consent (high-tech) PDF informed consent document.
  Interventions: Behavioral: Video consent (high-tech); Behavioral: PDF informed consent document
- Low-tech video consent (Experimental): Participants in this arm will be provided with informed consent information through viewing a "talking head" video produced by a non-professional presenter, with widely available and inexpensive video equipment. Intervention is "video consent (low-tech)", PDF informed consent document.
  Interventions: Behavioral: Video consent (low-tech); Behavioral: PDF informed consent document
- FAQ consent (Experimental): Participants in this arm will be provided with informed consent content through an interactive "frequently asked questions" format, in which the participant will click on a question and be shown text that provides an answer to that question. Major informed consent topics will have one or more question and answer pairs. Intervention is "FAQ format consent", PDF informed consent document
  Interventions: Behavioral: FAQ format consent; Behavioral: PDF informed consent document
- Standard consent process (Active Comparator): Participants in this arm will be provided with informed consent content by being shown a standard informed consent document in a scrolling window within the browser window, PDF informed consent document
  Interventions: Behavioral: Standard consent; Behavioral: PDF informed consent document

INTERVENTIONS:
Behavioral: Video consent (high-tech) — Consent provided by an animated video with captions
  Arms: Hi-tech video consent
Behavioral: Video consent (low-tech) — This consent is a video production of the informed consent information, taped using a staff member with basic video equipment.
  Arms: Low-tech video consent
Behavioral: FAQ format consent — This consent modality will present the basic information from the informed consent in an interactive, "frequently asked questions" format. Upon clicking each question, the participant will be shown a short text response to that question.
  Arms: FAQ consent
Behavioral: Standard consent — The standard consent form will present the full informed consent document in a scrolling text window within the browser window. Participants will be asked to review the document online.
  Arms: Standard consent process
Behavioral: PDF informed consent document — A PDF of the full consent document will be available for download, through hyperlink on the consent page. This is provided for video (low-tech), video (high-tech), FAQ format, and standard informed consent.

SUMMARY:
A two-part study to test the efficacy of alternative consent procedures and the efficacy of alternative methods to improve survey completion.

DETAILED DESCRIPTION:
Men who have sex with men are the risk population most heavily impacted by HIV in the United States by any measure; in 2009, at least 61% of new HIV infections were estimated to have occurred in MSM. MSM are experiencing an increase in HIV transmission that has been occurring since at least 1990, and accelerated in multiple North American and European countries from 2000-2005. The expansion of the HIV epidemic has been proposed to be attributable, in part, to the extent to which the internet has facilitated sexual connectivity among MSM.

Researchers have attempted to reach MSM for HIV prevention research and intervention on the internet. In the past 10 years, there has been a proliferation of internet surveys and HIV research studies among men who have sex with men that utilize the internet for data collection and, in some cases, the delivery of HIV prevention content. The development of internet-based interventions has been recently identified as especially promising because of its potential for scalability. However, there are also important limitations to internet-based data collections and prevention studies. The most important of these relate to representativeness and opportunities to introduce bias to data collections and differences in access to and use of internet among different subgroups of MSM. Equally important, although less discussed, are the unique ethical and human research protections challenges posed by online sexual health prevention studies.

The investigators will conduct a series of experiments that will result in improved knowledge of how to conduct internet-based HIV prevention research with MSM in ways that improve the protection of human subjects and decrease biases in data collections. The design will consist of preparatory online qualitative research with up to 100 MSM, followed by two cross-sectional randomized controlled trials of MSM recruited online; a total of 2440 MSM will be enrolled in the two randomized quantitative studies (1,440 in Study 1 to determine optimal methods to provide informed consent, online, and 1000 in Study 2 to determine how to best improve retention in online surveys). About 2440 men will be enrolled in the study in total. This summary describes Study 1; a separate submission will be completed for Study 2.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-34
* have had sex with another man in the past 12 months

Exclusion Criteria:

* female, transgender
* younger than 18 years old
* older than 34 years old
* have not had sex with a man in the past 12 months

Ages: 18 Years to 34 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2405 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Knowledge of Consent Information | At baseline (time zero)
  Correct knowledge of key aspects of the consent document will be operationalized by a count of the correctly answered consent recall items placed at the end of the survey, expressed as the number of correct items as a continuous measure.

SECONDARY OUTCOMES:
Proportion of eligible men who consent | Time of informed consent (baseline)
  The proportion of eligible men who consent to participate in the study; this secondary outcome is applicable only to the randomized study of alternative forms of informed consent administration.
Engagement with Consent Information | Time of consent
  We will measure engagement with the consent information by recording the amount of time a participant spends on the consent page before clicking to the first page of the survey.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick S Sullivan, PhD, Principal Investigator — Emory University
Locations (1):
- Rollins School of Public Health, Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Hall E, Sanchez T, Stephenson R, Stein AD, Sineath RC, Zlotorzynska M, Sullivan P. Randomised controlled trial of incentives to improve online survey completion among internet-using men who have sex with men. J Epidemiol Community Health. 2019 Feb;73(2):156-161. doi: 10.1136/jech-2018-211166. Epub 2018 Oct 31. PMID 30381466
- [Derived] Hall EW, Sanchez TH, Stein AD, Stephenson R, Zlotorzynska M, Sineath RC, Sullivan PS. Use of Videos Improves Informed Consent Comprehension in Web-Based Surveys Among Internet-Using Men Who Have Sex With Men: A Randomized Controlled Trial. J Med Internet Res. 2017 Mar 6;19(3):e64. doi: 10.2196/jmir.6710. PMID 28264794